CLINICAL TRIAL: NCT02416128
Title: Use of Topical Euphrasia, a Homeopathic Remedy in Ophthalmology
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Larkin Community Hospital (Other)
Collaborators: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: LCH-4-012015
Record Dates: First submitted 2015-03-26; First posted 2015-04-14 (Estimated); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Iritis
MeSH Terms: conditions — Iritis | interventions — euphrasiae herba; prednisolone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iritis prevention after LPI: prednisolone (Active Comparator): To use prednisolone acetate after and peripheral laser iridotomy to determine efficacy and side effects compared to arm 2.
  Interventions: Drug: Prednisolone acetate
- Iritis prevention after LPI: euphrasia (Experimental): To use euphrasia after and peripheral laser iridotomy to determine efficacy and side effects compared to arm 1.
  Interventions: Drug: Euphrasia

INTERVENTIONS:
Drug: Euphrasia — 1 drop in the treated eye QID X 10 days
  Other Names: Eyebright
  Arms: Iritis prevention after LPI: euphrasia
Drug: Prednisolone acetate — 1 drop in the treated eye QID X 10 days
  Other Names: Pred Forte
  Arms: Iritis prevention after LPI: prednisolone

SUMMARY:
The investigators plan to use an herbal eye drop, Euphrasia, aka Eyebright, for post-operative inflammation for Peripheral Laser Iridotomy for the treatment of narrow angle glaucoma. A peripheral Laser Iridotomy is a simple laser procedure with few complications if the patient follows the post-operative instructions. In this procedure, a blue-green Argon laser is used to create an orifice in the iris to open the angle by allowing the aqueous from behind the iris to enter the anterior chamber. Rarely the procedure needs to be repeated. The main complications from this surgery are postoperative inflammation, bleeding, and postoperative pressure spikes.

The investigators will be using Weleda's Euphrasia D3 eye drops. The investigators plan to do a double blinded randomized control trial to objectively measure ocular inflammation in the same process that was used for the steroid eye drops that are currently out on the market. Some patients will be receiving steroids, prednisolone acetate, others, the herbal eye drop.

DETAILED DESCRIPTION:
Status post Peripheral Laser Iridotomy Beraja Medical Institute has guidelines for the use of steroids after a Peripheral Laser Iridotomy. Patients are normally given prednisolone acetate ophthalmic solution, USP 1.0% to be used four times a day for seven days after the surgery. This protocol will also be used for the Euphrasia drops. This will help us compare the efficacy of the drugs as well as maintain a double blinded study.

Patients will be given blank bottles with only an ID number containing either prednisolone acetate or the Euphrasia eye drop. Bottles will be numbered sequentially by the Larkin Community Hospital pharmacy resident once the drops have been transferred by her and records of which bottles contain which drops will then be stored on the local intranet.

Patients will be given the exact same instructions as well as the instruction to come in/call the on-call resident immediately if there are any adverse side effects, and explained that the most common of which are expected to be signs of inflammation or allergy to the medication. The symptoms that the patients will be advised to call in for will be: redness, swelling, burning or itching lasting more than a few minutes, decrease/loss of vision lasting more than a few minutes. The phone number for the on-call resident is in the consent form. The patient will be given another copy of the consent form, if they do not have it, with the phone number of the on-call resident highlighted.

Patients will be followed up by a resident ophthalmologist on days eight and fifteen post-operatively to measure anterior chamber cell clearing and pain. The resident will only know which number bottle was used, not the drops in the bottleThe resident will also be measuring intraocular pressure, using a Goldman tonometer, and noting any other adverse effects or change in medication or dosing.Goldman tonometers are the most common way that an ophthalmologist checks a patient's intraocular pressure. It is done by using a topical anesthetic and dye instilled onto the cornea. The resident then places the Goldman tonometer onto the cornea, using a slit lamp, and measures the intraocular pressure. An attending ophthalmologist will recheck all findings and intervene, if necessary. These days and measures of efficacy are being used because these are the days and efficacy measures that were used to determine efficacy of multiple different steroid eye drops.

The goal of this project is to determine if Euphrasia eye drops are, at the very least, non-inferior to steroids in controlling intraocular inflammation in the post-operative period after peripheral laser iridotomy used in the treatment of narrow angle glaucoma. Euphrasia has been used for centuries for treating conjunctivitis, but there is no standardized method for delivery and very few other studies to prove its efficacy. Currently, steroid eye drops are the first choice to reduce intraocular inflammation. They are used after surgery, uveitis, and certain forms of conjunctivitis. The biggest problem with steroids is that some patients are "steroid responders." These individuals respond to the steroids by having a very large increase in their intraocular pressure which can lead to optic nerve damage. Up to 4% of patients who use steroids can have spikes in their pressures of up to 31mmHg, where normal intraocular pressure is 21 or less. These side effects can occur in as little of 5 days of taking the steroid eye drops. Other, less common side effects are: cataracts, exacerbation of bacterial/viral infections, ptosis, mydriasis, scleral melting, and eyelid skin atrophy.

With a recent shift in the American public to wanting to use herbal supplements and medications, it is very important to have clinical studies done to prove the efficacy of this herb. It is also important to be able to give the public a treatment that has been proven to work and is compounded safely and reproducibly.

There are two previous studies that were done in Germany, that have shown both the safety and efficacy of Euphrasia when used topically to treat inflammatory conditions of the eye (Stoss, M et.al. "Prospective Cohort Trial of Euphrasia Single-dose Eye Drops in Conjunctivitis." The Journal of Alternative and Complementary Medicine, Vol. 6, Number 6, 2000. pp499-508.) (Toelg, Michael. "Euphrasia D3 Eye Drops in Children." http://www.anthromed.org/Article.aspx?artpk=676 Accessed 2 July 2013.).

To achieve our goals, a comparison of the Euphrasia eye drop products that are currently on the market must be done. Weleda's Euphrasia D3 eye drops will be tested against prednisolone acetate eye drops to compare efficacy in reducing intraocular inflammation in the post-operative period after a peripheral laser iridotomy. This will be measured using a similar protocol used to show efficacy of steroidal eye drops already on the market. The investigator swill be measuring inflammation, intraocular pressure, and assessing pain at given intervals during the patient's post-operative period. The investigators will also be looking for specific signs of side effects that are known to occur with steroids and any other unwanted side effects, see research strategy for specifics.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Peripheral Laser Iridotomy

Exclusion Criteria:

* Patients who have had an allergic reaction to Euphrasia (this will be asked to the patient at time of )
* Patients who have had an adverse reaction to steroids (obtained by chart review to determine safety of drop use)
* Patients who have inflammation before the LPI (Noted by seeing cell in the anterior chamber)
* Patients who had any complications during their cataract surgery (obtained by chart review to determine safety of procedure)
* Patients in whom more than 1500mW of energy was used during the Peripheral Laser Iridotomy
* Patients in whom the laser was used more than 130 times during the Peripheral Laser Iridotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04-30 (Estimated); Primary Completion 2016-03-25 (Actual); Study Completion 2016-03-25 (Actual)

PRIMARY OUTCOMES:
Anti-inflammatory | 15 days post laser
  Quantitative amount of cell in the anterior chamber (0-5) Measurement of cell in the anterior chamber: 0 = 0 cells; 1 = 1 to 10 cells; 2 = 11 to 20 cells; 3 = 21 to 50 cells; and 4 = >50 cells (based on studies used to assess efficacy of other topical steroids)

SECONDARY OUTCOMES:
Side effects | 15 days post laser
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability
Pain prevention | 15 days post laser
  Pain assessment: Yes or No pain Pain will be measured as quantitative (Yes/No) (based on studies used to assess efficacy of other topical steroids)

CONTACTS AND LOCATIONS:
Overall Officials: Austin Bach, DO, Principal Investigator — Larkin Community Hospital/Nova Southeastern University

IPD SHARING:
Plan to Share IPD: No
Study was terminated

REFERENCES:
- [Result] ARMALY MF. EFFECT OF CORTICOSTEROIDS ON INTRAOCULAR PRESSURE AND FLUID DYNAMICS. I. THE EFFECT OF DEXAMETHASONE IN THE NORMAL EYE. Arch Ophthalmol. 1963 Oct;70:482-91. doi: 10.1001/archopht.1963.00960050484010. No abstract available. PMID 14078870
- [Result] BECKER B, MILLS DW. CORTICOSTEROIDS AND INTRAOCULAR PRESSURE. Arch Ophthalmol. 1963 Oct;70:500-7. doi: 10.1001/archopht.1963.00960050502012. No abstract available. PMID 14078872
- [Result] Foster CS, Forstot SL, Wilson LA. Mortality rate in rheumatoid arthritis patients developing necrotizing scleritis or peripheral ulcerative keratitis. Effects of systemic immunosuppression. Ophthalmology. 1984 Oct;91(10):1253-63. doi: 10.1016/s0161-6420(84)34160-4. PMID 6514289
- [Result] Stoss M, Michels C, Peter E, Beutke R, Gorter RW. Prospective cohort trial of Euphrasia single-dose eye drops in conjunctivitis. J Altern Complement Med. 2000 Dec;6(6):499-508. doi: 10.1089/acm.2000.6.499. PMID 11152054
- See also: Congdon NG, Schein OD, von Kulajta P, Lubomski LH, Gilbert D , Katz J. "Corneal Complications Associated with Topical Ophthalmic Use of Nonsteroidal Antiinflammatory Drugs." Journal of Cataract Refractive Surgery. 2001 ;27(4):622- 631. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC1359011/
- See also: Cullne, K., Golosinkiy, A. "Ambulatory Surgery in the United States, 2006." National Health Statistics Report Number 11, Revised September 4, 2009. — http://www.cdc.gov/nchs/data/nhsr/nhsr011.pdf
- See also: Shields MB. Textbook of Glaucoma. 4th ed. Philadelphia: Williams & Wilkins; 2000 . — http://www.alibris.com/Textbook-of-Glaucoma-M-Bruce-Shields/book/6630168
- See also: SBL's Euphrasia 10% Eye Drops — https://sblglobal.com/home
- See also: Toelg, Michael. "Euphrasia D3 Eye Drops in Children." — https://www.anthromed.org/library/2019/1/4/euphrasia-d3-eye-drops-in-children?rq=Euphrasia%20D3%20Eye%20Drops%20in%20Children
- See also: White, L., Foster, S. The Herbal Drugstore. Penguin Group, 2002. — http://www.barnesandnoble.com/w/the-herbal-drugstore-linda-b-white/1013440593?ean=9780451205100